CLINICAL TRIAL: NCT04553081
Title: Virological and Immunological Assessment in HIV Positive Participants on 2DR Versus 3DR in a Prospective Randomized Controlled Switch Trial
Brief Title: 2DR Versus 3DR in a Prospective Randomized Controlled Switch Trial
Acronym: 2DR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-7052
Record Dates: First submitted 2020-05-29; First posted 2020-09-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: HIV-1-infection
Keywords: HIV; dual therapy; triple therapy; virological control; immune activation; metabolic complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dovato (Active Comparator): We aim to include 134 adult HIV-infected patients with HIV RNA < 50 copies/mL for at least 3 months on any stable 2nd generation integrase based triple therapy antiretroviral regimen. Patients will be randomized 1:2 to switch to or stay on the triple regimen BIC/TAF/FTC (Biktarvy) (N=45) or to switch to the dual regimen DTG/3TC (Dovato) (N=89).
  Interventions: Drug: Dual versus triple therapy in treatment of HIV-1 infection.
- Biktarvy (Active Comparator): We aim to include 134 adult HIV-infected patients with HIV RNA < 50 copies/mL for at least 3 months on any stable 2nd generation integrase based triple therapy antiretroviral regimen. Patients will be randomized 1:2 to switch to or stay on the triple regimen BIC/TAF/FTC (Biktarvy) (N=45) or to switch to the dual regimen DTG/3TC (Dovato) (N=89).
  Interventions: Drug: Dual versus triple therapy in treatment of HIV-1 infection.

INTERVENTIONS:
Drug: Dual versus triple therapy in treatment of HIV-1 infection. — cfr arm description
  Other Names: not applicatble

SUMMARY:
The aim of this study is to monitor virological and immunological markers in participants who are switching from a classic triple drug regimen (3DR) to dual therapy (2DR). We aim to monitor whether this has an influence on different parameters such as severity of HIV disease (evaluated by viral load and viral reservoir size), presence of non-AIDS related health complications, impact the phenotype and function of the immune system.

By conducting this study we want to assess whether switching from 3DR to 2DR implies an increased risk for 'subclinical' failure. We especially want to make sure that this switch does not increase the HIV reservoir, does not increase inflammation or immune exhaustion in patients living with HIV and that it can be considered as a safe long term alternative for the classic 3DR.

The primary objective is to demonstrate non inferiority at W48 of the 2DR DTG/3TC (Dovato) regimen compared to BIC/TAF/FTC (Biktarvy) in terms of the amount of intact replication competent HIV sequences with a non-inferiority margin of 12% quantified by the fraction intact HIV viral sequences quantified by an intact proviral DNA assay, present in blood CD4 cells.

DETAILED DESCRIPTION:
In HIV care we have been facing a paradigm change over the last years, reaching an ultimatum with the reimbursement of a 2DR regimen both in naïve as in switch patients.

The rationale behind dual therapy is interesting, namely lower cost, less side-effects, more preserved treatment options, less interactions.

However, from a patient and clinician's perspective this requires a paradigm change after an era of successful treating patient with 3DR.

In the past 2DR and even 1DR treatments have been proposed as an alternative for 3DR, however results were often disappointing and these regimens were only suitable for a selection of patients, often requiring intensification of follow-up.

Recently dual therapy with integrase inhibitor dolutegravir has shown very promising results both in switch (TANGO study) with no virological failure related to this regimen over 48 weeks and in naïve patients (GEMINI study) with no resistance mutations at 96 weeks. Moreover, time to undectability was statistically not different from the 3DR group and the small amount of data available on in depth analysis of the reservoir and immunological parameters were reassuring.

Comparative data however on immunological and virological parameters are lacking therefore we want to conduct the present clinical trial to further elaborate on this important question.

Recent data show that newer ARVs, among which integrase inhibitors and TAF, are associated with weight gain. Further data is required to investigate the patterns of weight change with these ARVs and any associated metabolic impact.

So far, DTG/3TC has been assessed in 3 phase III clinical trials: GEMINI-1, GEMINI-2 and TANGO. GEMINI-1 and GEMINI-2 are two large identically designed phase 3 studies that compare the 2DR DTG+3TC once daily with a first-line recommended 3DR DTG + 2 nucleoside reverse transcriptase inhibitors (NRTIs) (tenofovir disoproxil (TDF)/FTC) once daily in treatment-naïve People living with HIV (PLHIV) (Cahn 2019). The primary objective of TANGO is to demonstrate the non-inferior antiviral activity of switching to DTG+3TC once daily compared to the continuation of TAF-based regimens (TBR) over 48 weeks in ART-experienced, virologically suppressed PLHIV (Van Wyk 2020). The primary results of these trials have been published (Cahn 2019, Van Wyk 2020) while the trials continue in order to collect longer-term data.

GEMINI-1 and GEMINI-2 are 2 twin phase 3, randomised, double-blind, active-controlled, multicentre, parallel-group, noninferiority studies conducted in treatment-naive patients with HIV-1 RNA of 1000 to ≤500,000 c/mL at screening. Patients are randomised 1:1 to receive DTG+3TC once daily or DTG plus FDC tablet of TDF/FTC once daily. The results of GEMINI-1, GEMINI-2, and the pooled analysis demonstrated that DTG+3TC has a high level of efficacy and safety and is noninferior to 3DR DTG+TDF/FTC. In the pooled analysis, 91% of patients in the DTG+3TC arm and 93% of patients in the DTG+TDF/FTC arm achieved plasma HIV-1 RNA <50 c/mL by Week 48. The Week 96 secondary efficacy analysis demonstrated that DTG+3TC continued to provide a high level of clinical efficacy. A similar proportion of subjects in each treatment group achieved the secondary efficacy endpoint of plasma HIV-1 RNA <50 c/mL at Week 96 for GEMINI-2 and pooled analysis. Based on the Food and drug administration (FDA) Snapshot algorithm, DTG+3TC is noninferior to DTG+TDF/FTC in the individual studies as well as the pooled analysis at Week 48 and at Week 96. The subgroup analyses further supported the noninferiority of DTG+3TC at both Week 48 and Week 96. Moreover, few patients experienced CVW by Week 48, with comparable rates across treatment arms (<1% in each) and fewer AEs were observed in the DTG+3TC arm compared to DTG+TDF/FTC. No treatment-emergent resistance mutation were observed in these patients up to Week 96, demonstrating DTG+3TC's high barrier to resistance. The incidence of drug-related AEs at Week 48 in the DTG+3TC arm was low (126/716; 18%) and lower than that in the DTG+TDF/FTC arm (169/717; 24%). The most common (≥1%) drug-related Grade 2-4 AE in both arms was headache (1% in both arms). Low rates of drug-related AEs were also observed at Week 96 for both arms, with slightly more but comparable overall AEs and slightly more drug-related AEs in the DTG+TDF/FTC arm compared with the DTG+3TC arm.

TANGO is a 200-week, phase 3, randomised, open-label, active-controlled, multicentre, parallel-group study to assess the noninferior antiviral activity and safety of replacing a TBR with a 2DR of DTG+3TC in HIV-infected adults who are virologically suppressed and stable on TBR (Van Wyk 2020). The results of TANGO demonstrate that DTG+3TC has a high level of efficacy and safety for patients switching from TBR. Based on the FDA Snapshot virologic failure, DTG+3TC is noninferior to TBR at Week 24 (Ait-Khaled 2019, Van Wyk 2020). Very few (<1%) patients experienced virologic failure in both treatment arms. Only one patient in the TBR arm had a CVW by Week 24. A greater proportion of patients in the DTG+3TC arm experienced Serious Adverse Events (SAEs) (but not drug-related SAEs), drug-related adverse events (AEs), and AEs leading to withdrawal from the study compared with the TBR arm in the first 24 weeks of the study as expected due to the switch study design.

The various clinical trials ongoing and planned for DTG/3TC are further supported by real-world evidence. These real-world studies have findings consistent with the results observed in clinical trials.

The primary objective is to demonstrate non inferiority at W48 of the 2DR DTG/3TC (Dovato) regimen compared to BIC/TAF/FTC (Biktarvy) in HIV-1 infected individuals in terms of the amount of intact replication-competent HIV-1 sequences with a non-inferiority margin of 12% quantified by the fraction intact HIV viral sequences quantified by IPDA, present in blood CD4 cells.

1. Quantification of immune activation markers in both arms, will be explored as secondary objective and should not differ more than 20%. The power calculation is however calculated based on the primary objective.

   Assessment at baseline, W48 and W144.
   * Inflammation markers: IL-6, hs-CRP (of CRP) (other: IL_8, IP10, TNF, B2M, CXCL1, IL21, Hyaluric acid)
   * Markers of coagulopathy: D-Dimers
   * T cell activation markers: HLA-DR, CD38 on both CD4 and CD8; soluble markers: sCD27, sCH40 ligand
   * T cell exhaustion markers: PD-1, CD28, CD57
   * Markers of microbial translocation: sCD14
   * CD4/CD8 ratio
2. In addition, the secondary objective is to assess impact of the DTG/3TC vs BIC/FTC/TAF on metabolic health. Therefore, as secondary endpoint metabolic health will be assessed through incidence of metabolic syndrome, weight/BMI change, waist circumference, and insulin resistance. Finally, dual-energy x-ray absorptiometry (DXA) scans will be performed to assess body composition and fat distribution and bone mineral density and FibroScans will be performed to assess liver steatosis and fibrosis.
3. As a third secondary objective we will assess the impact of switching through a patient questionnaire.
4. The fourth secondary objective is to demonstrate non inferiority at W144 of the 2DR DTG/3TC (Dovato) regimen compared to BIC/TAF/FTC (Biktarvy) in HIV-1 infected individuals in terms of the amount of intact replication-competent HIV-1 sequences with a non-inferiority margin of 12% quantified by the fraction intact HIV viral sequences quantified by IPDA, present in blood CD4 cells.

ELIGIBILITY:
Inclusion Criteria:

* Age = or >18 years.
* Ability and willingness to provide written informed consent.
* Ability to attend the complete schedule of assessments and patient visits.
* Ability and willingness to have blood samples collected and stored indefinitely and used for various research purposes.
* HIV RNA < 50 copies/mL for at least 3 months on a 2nd generation INSTI based regimen.
* Females of childbearing potential should be on effective contraception

Exclusion Criteria:

* Current presence of opportunistic infection (AIDS defining events as defined in category C of the CDC clinical classification).
* Evidence of active HBV infection (Hepatitis B surface antigen positive or HBV viral load positive in the past and no evidence of subsequent seroconversion (seroconversion= HBV antigen or viral load negative and positive HBV surface antibody).
* Evidence of active HCV infection: HCV antibody positive result within 60 days prior to study entry with positive HCV viral load or, if the HCV antibody result is negative, a positive HCV RNA result within 60 days prior to study entry.
* Pregnancy or breastfeeding.
* Patients unable to understand the study protocol or any other condition that in the investigator's opinion may compromise compliance with the study protocol
* Decompensated liver cirrhosis (Child-Pugh B/C)
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (apart from hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones)
* Psychiatric and psychological disorders, which in the opinion of the investigator, will interfere with the trial conduct or safety of the participant.
* Previous participation in a trial evaluating an immune modulating agent.
* Active drug or alcohol use/addiction such that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Treatment failure on an integrase inhibitor containing regimen and reported baseline resistance
* Creatinine Clearance <50
* Tuberculosis treatment
* Documented M184V
* Previous virological failure >200 copies/mL on NRTI
* Subjects with history or presence of allergy to any of the study drugs or their components
* ALT >5 times the ULN, OR ALT >3xULN and bilirubin >1.5xULN (with >35% direct bilirubin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Difference in amount of intact replication-competent HIV-1 sequences in CD4 cells between 2 regimens | 48 weeks
  The primary objective is to demonstrate non inferiority at W48 of the 2DR DTG/3TC (Dovato) regimen compared to BIC/TAF/FTC (Biktarvy) in HIV-1 infected individuals in terms of the amount of intact replication-competent HIV-1 sequences with a non-inferiority margin of 12% quantified by the fraction intact HIV viral sequences quantified by the intact proviral DNA assay (IPDA), present in blood CD4 cells.

SECONDARY OUTCOMES:
Full length sequencing of the virus | 240 weeks
  Full length sequencing of the virus at baseline, W48, W144 and W240
Quantification of interleukin-6 (IL-6) | 240 weeks
  Quantification of IL-6 at baseline, W48, W144 and W240
Quantification of high-sensitivity C-reactive protein (hs-CRP) | 240 weeks
  Quantification of hs-CRP at baseline, W48, W144 and W240
Quantification of D-Dimers | 240 weeks
  Quantification of D-Dimers at baseline, W48, W144 and W240
Quantification of Human Leukocyte Antigen - DR isotype (HLA-DR) | 240 weeks
  Quantification of HLA-DR at baseline, W48, W144 and W240
Quantification of cluster of differentiation 38 (CD38) | 240 weeks
  Quantification of CD38 on both cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) immune cells at baseline, W48, W144 and W240
Quantification of soluble cluster of differentiation 27 (sCD27) | 240 weeks
  Quantification of sCD27 at baseline, W48, W144 and W240
Quantification of soluble cluster of differentiation 40 (sCD40) | 240 weeks
  Quantification of sCD40 at baseline, W48, W144 and W240
Quantification of programmed cell death protein 1 (PD-1) | 240 weeks
  Quantification of the T cell exhaustion marker PD-1 at baseline, W48, W144 and W240
Quantification of cluster of differentiation 28 (CD28) | 240 weeks
  Quantification of the T cell exhaustion marker CD28 at baseline, W48, W144 and W240
Quantification of cluster of differentiation 57 (CD57) | 240 weeks
  Quantification of the T cell exhaustion marker CD57 at baseline, W48, W144 and W240
Quantification of soluble cluster of differentiation 14 (sCD14) | 240 weeks
  Quantification of markers of microbial translocation sCD14 at baseline, W48, W144 and W240
Quantification of CD4/CD8 ratio | 240 weeks
  Quantification of CD4/CD8 ratio at baseline, W48, W144 and W240
Incidence of metabolic syndrome | 240 weeks
  Metabolic health will be assessed through incidence of metabolic syndrome at baseline, W48, W144 and W240
Weight/body mass index (BMI) change | 240 weeks
  Metabolic health will be assessed through weight/BMI change at baseline, W48, W144 and W240
Waist circumference | 240 weeks
  Metabolic health will be assessed through waist circumference at baseline, W48, W144 and W240
Insuline resistance | 240 weeks
  Metabolic health will be assessed through insuline resistance at baseline, W48, W144 and W240
Dual-energy x-ray absorptiometry (DXA) | 240 weeks
  Bone mineral density will be assessed through DXA at baseline, W48, W144 and W240
FibroScans | 240 weeks
  Fat distribution will be assessed through FibroScans at baseline, W48, W144 and W240
Switch questionnaire | 240 weeks
  The impact of switching will be assessed through a patient switch questionnaire at baseline, W48, W144 and W240
Duplex carotis | 240 weeks
  In all participants or in a subgroup identified as high and very high cardiovascular risk group will be proposed a duplex carotis at W240 to assess the intima media tickness as a surrogate marker for generalised atherosclerosis and risk of cardio-vascular disease.
Quantification of lipoproteine A | 168 weeks
  Quantification of lipoproteine A at W168

CONTACTS AND LOCATIONS:
Overall Officials: Linos Vandekerckhove, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delporte M, Lambrechts L, Blomme EE, van Snippenberg W, Rutsaert S, Verschoore M, De Smet E, Noppe Y, De Langhe N, De Scheerder MA, Gerlo S, Vandekerckhove L, Trypsteen W. Integrative Assessment of Total and Intact HIV-1 Reservoir by a 5-Region Multiplexed Rainbow DNA Digital PCR Assay. Clin Chem. 2025 Jan 3;71(1):203-214. doi: 10.1093/clinchem/hvae192. PMID 39749517
- [Derived] De Scheerder MA, Degroote S, Delporte M, Kiselinova M, Trypsteen W, Vincke L, De Smet E, Van Den Eeckhout B, Schrooyen L, Verschoore M, Muccini C, Vanherrewege S, Caluwe E, De Buyser S, Gerlo S, Blomme E, Vandekerckhove L. In-depth Analysis of the HIV Reservoir Confirms Effectiveness and Safety of Dolutegravir/Lamivudine in a Phase 4 Randomized Controlled Switch Trial (RUMBA). J Infect Dis. 2025 Feb 4;231(1):e91-e100. doi: 10.1093/infdis/jiae405. PMID 39226296